CLINICAL TRIAL: NCT00823238
Title: Comparison of Antibiotics for Pseudomonas in Early CF
Acronym: CAPEC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Terry L. Noah, MD, UNC Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCRC2197
Record Dates: First submitted 2008-12-29; First posted 2009-01-15 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2011-04

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Ceftazidime; Tobramycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- systemic (Active Comparator)
  Interventions: Drug: ceftazidime and tobramycin
- inhaled (Active Comparator)
  Interventions: Drug: inhaled tobramycin

INTERVENTIONS:
Drug: ceftazidime and tobramycin
  Arms: systemic
Drug: inhaled tobramycin
  Arms: inhaled

SUMMARY:
This is a prospective, randomized clinical trial comparing the effects of these 2 modes of antibiotic treatment on BALF inflammation in young, P. aeruginosa-positive CF patients.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is a genetic disorder which is typically fatal during early adulthood, due to progressive bronchiectasis and respiratory failure. Chronic lung infection with Pseudomonas aeruginosa begins in early life and is clearly associated with decline (especially mucoid phenotypes), making this infection a major target of therapy. The inflammatory response to infection may also be dysregulated in CF, so that suppression of airway inflammation is a second major goal of therapy. However, "best practice" for treatment of Pseudomonas infection in early CF is not defined (several recently published commentaries available upon request) and is a critical issue currently in clinical management of CF. Inhaled tobramycin alone has been reported to be effective at short-term eradication of P. aeruginosa from bronchoalveolar lavage fluid (BALF) in children with cystic fibrosis (CF) age 3 mo-6 yr, but inflammation was unaffected by this treatment, and recurrence of infection occurred fairly quickly for mucoid strains. The ideal treatment would result in long-term reduction in both bacterial quantity and inflammation. Some bacteria in the CF airway may be both inaccessible to inhaled antibiotics, and "hidden" from BALF, by location in inspissated secretions, and P. aeruginosa may not be effectively eradicated in paranasal sinuses. Thus, it is reasonable to hypothesize that treatment with parenteral antibiotics provides better overall eradication of organisms and consequently reduced stimulus for ongoing or recurrent inflammation in the airways. We therefore propose a prospective, randomized clinical trial comparing the effects of these 2 modes of antibiotic treatment on BALF inflammation in young, P. aeruginosa-positive CF patients.

ELIGIBILITY:
Inclusion Criteria:

1. Positive respiratory culture (sputum, BALF, or deep pharyngeal culture) in the past 3 months for P. aeruginosa. Those who are culture positive for both P. aeruginosa and additional bacteria (S. aureus, H. influenzae) would also be eligible (but see microbiologic exclusions below). Children with either first isolate or chronic/repeated P. aeruginosa infection are eligible.
2. Clinically stable as defined by:

   1. No systemic anti-P. aeruginosa antibiotics in the past 2 mo, and no TOBI in the past 1 month;
   2. No pulmonary exacerbation in the past 1 mo (definition furnished on request); and
   3. FEV1 ≥ 70% predicted (best baseline past 6 months and at study entry) for those old enough to reliably test spirometric lung function.

Exclusion Criteria:

1. Recent (within past 2 mo) use of systemic anti-Pseudomonas antibiotics, with the exception of chronic (three times a week) azithromycin;
2. Recent (within past 2 wk) use of systemic anti-inflammatory agents;
3. Mycobacterial pathogens on AFB smear at initial bronchoscopy;
4. Multiple-drug resistant (MDR)-P. aeruginosa, or oxacillin-resistant S. aureus (ORSA) on respiratory cultures in the past 3 months. If either MDR-P. aeruginosa, or ORSA are isolated at the initial bronchoscopy, subjects will be excluded and results discussed with primary caregiver.
5. Viral pathogens are occasionally isolated from BALF but this may take 2-3 weeks. Thus, any subjects with this result after initial bronchoscopy will likely have completed the treatment protocol, but would not undergo bronchoscopy #2.
6. History of reactions to or problems with anesthesia or sedation.
7. History of reactions to or problems with aminoglycosides (medicines like tobramycin or gentamicin).
8. History of hemoptysis (coughing up blood) within 30 days prior to entry.
9. History of anemia or thrombocytopenia.
10. Administration of any investigational drug within 30 days prior to entry.
11. History of abnormal kidney function (greater than 1.5 times the upper limit of normal serum creatinine for age).
12. History of documented chronic hearing loss.
13. for children under the age of 3 months, prematurity defined as gestational age < 36 weeks.

Ages: 3 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2004-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terry Noah, MD, Principal Investigator — UNC-CH